CLINICAL TRIAL: NCT00347893
Title: Clinical Results of Selective Laser Trabeculoplasty in Treatment of Open Angle Glaucoma
Brief Title: The Efficacy of Selective Laser Trabeculoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glaucoma Research & Education Group (Other)
Collaborators: PharmaLogic Development, Inc. (Industry)
Other Study IDs: 22222
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension; Pseudo-Exfoliative Glaucoma; Pigment Dispersion Glaucoma
Keywords: Primary open angle glaucoma; Ocular hypertension; Pseudo-exfoliative glaucoma; Pigment Dispersion glaucoma; selective laser trabeculoplasty; intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Selective laser trabeculoplasty

SUMMARY:
Selective laser trabeculoplasty (SLT) is a new method to reduce intraocular pressure in eyes with open angle glaucoma or ocular hypertension. SLT may also be effective for cases with previously failed ALT procedures. We will study the efficacy and safety of the SLT procedure.

DETAILED DESCRIPTION:
Selective laser trabeculoplasty (SLT) has been shown to be a safe, well tolerated, and effective intraocular pressure reduction therapy for several forms of open-angle glaucoma. SLT produces significantly less disturbance to the trabecular meshwork and is theoretically more repeatable than the ALT procedure. This retrospective research will begin with cases treated in 2001. It will evaluate whether SLT is effective for patients who have had prior treatment with ALT and it will determine whether the IOP lowering effect is sustainable over time. It will also assess the efficacy of repeated SLT procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary open angle glaucoma, ocular hypertension, pseudo exfoliative glaucoma, pigment dispersion glaucoma

Exclusion Criteria:

* History of prior invasive glaucoma surgery

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G. Iwach, M.D., Principal Investigator — Glaucoma Research & Education Group
Locations (1):
- Glaucoma Center of San Francisco, San Francisco, California, United States